CLINICAL TRIAL: NCT04397523
Title: Use of COVID-19 Convalescent Plasma in the Patients Infected With COVID-19 (SARS-CoV-2) - Efficacy and Safety
Brief Title: Efficacy and Safety of COVID-19 Convalescent Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Transfusion Medicine of RNM (Other Government)
Collaborators: University Clinic for Infectious Diseases, North Macedonia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITM05/2020MKD
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Convalescent Plasma; COVID-19; SARS-CoV 2
Keywords: COVID-19; anti SARS-CoV-2 convalescent plasma; COVID-19 convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospitalized patients with SARS CoV-2 infection (Other): Hospitalized patients with SARS CoV-2 infection will receive an anti SARS-CoV-2 convalescent plasma
  Interventions: Biological: anti-SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: anti-SARS-CoV-2 convalescent plasma — Administration of convalescent plasma obtained from donors with prior documented SARS-CoV-2 infection

SUMMARY:
Administration of convalescent plasma obtained from donors with prior documented SARS-CoV-2 infection

DETAILED DESCRIPTION:
There are currently no proven therapeutic options for coronavirus disease (COVID-19), the infection caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Human convalescent plasma is an option for treatment of COVID-19. Experience from prior outbreaks with other coronaviruses, such as SARS-CoV-1, MERS and H1N1 shows that convalescent plasma can be effective. Convalescent plasma will be obtained by plasmapheresis or regular whole blood donation in subjects who recovered from COVID-19 and who are otherwise eligible for donation according to the Institutional protocol. Recipients will be COVID-19 patients requiring hospitalization. A blood-type matched transfusion of convalescent plasma will be infused and recipients will be followed up.

ELIGIBILITY:
Inclusion Criteria

Blood donors:

1. Age: >18 and <60 years
2. Body weight : >55 kg
3. Confirmed previous SARS CoV-2 infection
4. Minimum 28 days after the last symptom or finishing of the isolation, or
5. 21 day without symptoms from the date of the negative SARS CoV-2 test
6. Written informed consent to participate in this clinical trial, to donate plasma and to store the specimen for future testing.
7. Concentration of COVID-19 IgG antibodies more than 5 AU/ml (Because measurement of neutralizing antibody titers is not available now, storing of retention sample from the convalescent plasma donation is performed for determining antibody titers at a later date)
8. Male donors, or female donors who have not been pregnant, or female donors who have been pregnant tested negative for HLA antibodies
9. Individuals who meet all regular voluntary donor eligibility requirements

Patients/recipients:

1. Age: >18 years
2. Admitted to an acute care facility for the treatment of COVID-19 complications
3. Patients with severe or immediately life-threatening COVID-19, or
4. Patients who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening disease.
5. Informed consent provided by the patient or healthcare proxy

Exclusion Criteria:

Blood donors:

1. Age : <18 or >60 years
2. Female subjects who are pregnant
3. HIV1,2 hepatitis B,C or syphilis infection
4. Donors ineligible for regular voluntary blood donation

Patients/recipients:

1. Age : <18 years
2. Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products)
3. Patients who received in the past 30 days immunoglobulin therapy
4. Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rada Grubovic Rastvorceva, MD MSci PhD, Principal Investigator — Institute for Transfusion Medicine of RNM; Sedulla Useini, MD, Principal Investigator — Institute for Transfusion Medicine of RNM
Locations (1):
- Institute for Transfusion Medicine of RNM, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on request to other clinical researchers involved in similar trials or meta-analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Since the publication of results for the next 5 years
Access Criteria: Interested researchers should write to the principal investigators of this trial explaining why they need this data

REFERENCES:
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Huaxia, (2020). 'China puts 245 COVID-19 patients on convalescent plasma therapy', Xinhua.net, 2 February. Available at: http://www.xinhuanet.com/english/2020-02/28/c_138828177.htm
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Roback JD, Guarner J. Convalescent Plasma to Treat COVID-19: Possibilities and Challenges. JAMA. 2020 Apr 28;323(16):1561-1562. doi: 10.1001/jama.2020.4940. No abstract available. PMID 32219429
- [Background] https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-deviceexemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds Accessed on March 30,2020
- [Background] Guidance on collection, testing, processing, storage, distribution and monitored use. An EU programme of COVID-19 convalescent plasma collection and transfusion. EUROPEAN COMMISSION DIRECTORATE-GENERAL FOR HEALTH AND FOOD SAFETY, 08 April, 2020
- [Background] AABB's CCP Collection Protocol - Donor Eligibility, Processing, Labeling and Distribution, 03 April, 2020 http://www.aabb.org/advocacy/regulatorygovernment/Documents/COVID-19-Convalescent-Plasma-Collection.pdf
- [Derived] Grubovic Rastvorceva RM, Useini S, Stevanovic M, Demiri I, Petkovic E, Franchini M, Focosi D. Efficacy and Safety of COVID-19 Convalescent Plasma in Hospitalized Patients-An Open-Label Phase II Clinical Trial. Life (Basel). 2022 Oct 9;12(10):1565. doi: 10.3390/life12101565. PMID 36295001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Started | 200
Completed | 189
Not Completed | 11
Not completed — Lost to Follow-up | 3
Not completed — Transfer from/to other hospital | 8

BASELINE CHARACTERISTICS:
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.8)
Age, Customized [Count of Participants; unit: Participants]
  18-35 years | 11
  36-45 years | 23
  46-55 years | 47
  56-65 years | 56
  66-75 years | 41
  more than 75 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Macedonians | 139
  Ethnicity: Albanians | 36
  Ethnicity: others | 14
Region of Enrollment [Count of Participants; unit: Participants]
  North Macedonia | 189
Body Mass Index [Count of Participants; unit: Participants]
  18.5-24.9 kg/m^2 (normal) | 37
  25-29.9 kg/m^2 (overweight) | 95
  equal or more than 30 kg/m^2 (obese) | 57
ABO blood type [Count of Participants; unit: Participants]
  A | 94
  B | 32
  O | 47
  AB | 16
WHO progression score [Count of Participants; unit: Participants]
  WHO disease progression score 3 - hospitalized patients without oxygen support | 65
  WHO progression score 4 - hospitalized patients with oxygen support (nasal canila, oxygen mask) | 65
  WHO progression score 5 - hospitalized with high-flow oxygen support (noninvasive ventilation) | 59
Comorbidities [Count of Participants; unit: Participants]
  yes | 134
  no | 55
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Oxygenation Support
Description: The total number of days patients required respiratory support.
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Population: This is the number of patients that required respiratory support before CCP transfusion
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 124
days | 7.4 (5.2)

2. Primary Outcome: Hospital Length of Stay (LOS)
Description: Total number of days patients were admitted to the hospital after convalescent plasma transfusion.
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Population: The bellow are shown subgroups of participants according to the WHO disease progression scores 3,4 and 5, which all together comprises total investigated group of 189 participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
days
  total investigated group | 11.0 (5.3)
  patients with WHO disease progression score 3, which are not on oxygen support: number analyzed (Participants) | 65
  patients with WHO disease progression score 3, which are not on oxygen support | 8.6 (2.7)
  patients with WHO score 4, which are on oxygen support with nasal canila or oxygen mask: number analyzed (Participants) | 65
  patients with WHO score 4, which are on oxygen support with nasal canila or oxygen mask | 11.1 (4.7)
  patients with WHO score 5, which are on oxygen support with noninvasive ventilation: number analyzed (Participants) | 59
  patients with WHO score 5, which are on oxygen support with noninvasive ventilation | 13.6 (6.7)
Statistical Analysis 1: Comparison: Hospitalized Patients With SARS CoV-2 Infection; Test type: Other; p = 0.05, ANOVA — p=0.00000; df 2

3. Primary Outcome: ICU Admission
Description: Total number of subjects to be admitted to the ICU after the convalescent plasma transfusion.
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
Participants | 1

4. Primary Outcome: Number of Participants With Oxygenation Free Days
Description: Number of participants without oxygenation support after receiving convalescent plasma
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
Participants
  Participants with oxygenation free days before CCP transfusion | 65
  Participants with oxygenation free days 24 hours after CCP transfusion | 76
  Participants with oxygenation free days after 7 days after transfusion | 103
  Participants with oxygenation free days at discharge | 167

5. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with serious adverse events during the study protocol
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Groups:
- Hospitalized Patients With SARS CoV-2 Infection: Hospitalized adult patients with confirmed SARS CoV-2 infection will receive an anti SARS-CoV-2 convalescent plasma
  anti-SARS-CoV-2 convalescent plasma: Administration of convalescent plasma obtained from donors with prior documented SARS-CoV-2 infection
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
Participants | 0

6. Secondary Outcome: Type of Respiratory Support
Description: Type of supplemental oxygen support (e.g. nasal canula, high flow nasal canula, noninvasive ventilation, intubation and invasive mechanical ventilation, rescue ventilation)
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
Participants
  Nasal canula, oxygen mask before CCP transfusion | 65
  Nasal canula, oxygen mask 24 hours after CCP transfusion | 56
  Nasal canula, oxygen mask 7 days after CCP transfusion | 35
  Noninvasive ventilation, high flow nasal canula before CCP transfusion | 59
  Noninvasive ventilation, high flow nasal canula 24 hours after CCP transfusion | 56
  Noninvasive ventilation, high flow nasal canula 7 days after CCP transfusion | 25
  Intubation or invasive mechanical ventilation, before CCP transfusion | 0
  Intubation or invasive mechanical ventilation, 24 hours after CCP transfusion | 1
  Intubation or invasive mechanical ventilation, 7 days after CCP transfusion | 1
  Rescue ventilation before CCP transfusion | 0
  Rescue ventilation 24 hours after CCP transfusion | 0
  Rescue ventilation 7 days after CCP transfusion | 1

7. Secondary Outcome: Number of Participants With Different Clinical Outcomes Including Death, Critical Illness and Recovery
Description: Number of participants with different clinical outcomes including death, critical illness, limitation of activities and recovery
Time Frame: 28 days after transfusion or until hospital discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
Number analyzed (Participants) | 189
Participants
  total recovery | 164
  recovery with limitation of activities | 3
  death | 22
Statistical Analysis 1: Comparison: Hospitalized Patients With SARS CoV-2 Infection; Overall survival between the three WHO score groups 3, 4 and 5; Test type: Other; p = 0.05, Chi-squared — Chi- square = 24.98174, p = 0.00000; df = 2
Statistical Analysis 2: Comparison: Hospitalized Patients With SARS CoV-2 Infection; Correlation of mortality versus WHO disease progression score of patients; Test type: Other; p = 0.05, Chi-squared — p=0.000; df = 2
Statistical Analysis 3: Comparison: Hospitalized Patients With SARS CoV-2 Infection; Correlation of mortality versus stay in the intensive care unit (ICU); Test type: Other; p = 0.05, Chi-squared — p = 0.000; df = 1

ADVERSE EVENTS:
Time Frame: During hospitalization, after receiving convalescent plasma
Arm/Group | Hospitalized Patients With SARS CoV-2 Infection
All-Cause Mortality (participants affected / at risk) | 22/189
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 1/189
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hospitalized Patients With SARS CoV-2 Infection (N=189)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — rash on the skin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT04397523/Prot_SAP_000.pdf